CLINICAL TRIAL: NCT02979639
Title: Study to Evaluate the Impact of Reactogenicity on Quality of Life (QoL), After Administration of GSK Biologicals' Candidate Herpes Zoster Subunit (HZ/su) Vaccine (GSK1437173A) in Adults ≥ 50 Years of Age
Brief Title: Study to Evaluate the Impact of Reactogenicity on Quality of Life (QoL), After Administration of GlaxoSmithKline (GSK) Biologicals' Candidate Herpes Zoster Subunit (HZ/su) Vaccine (GSK1437173A) in Adults ≥ 50 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 204928
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster; Reactogenicity; Quality of life; Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK1437173A Group (Experimental): Subjects ≥ 50 years of age who will receive two doses of the GSK1437173A vaccine (first dose given at Month 0 and second dose given 2 months later) in this study.
  Interventions: Biological: GSK Biologicals Herpes Zoster subunit (HZ/su) vaccine (GSK 1437173A)

INTERVENTIONS:
Biological: GSK Biologicals Herpes Zoster subunit (HZ/su) vaccine (GSK 1437173A) — 2 doses administered by intramuscular (IM) injection into the deltoid muscle of the non-dominant arm on a 2 month schedule.

SUMMARY:
The purpose of this study is to evaluate the impact of reactogenicity of GSK Biologicals' HZ/su vaccine on Quality of Life (QoL) in adults ≥ 50 years of age

DETAILED DESCRIPTION:
The study will evaluate the impact of HZ/su vaccination on the QoL, 400 adults ≥ 50 years of age (YOA). Subjects will be asked to respond to a series of SF-36 and EQ-5D questionnaires before and after vaccination following a 2 month schedule. To estimate the impact of reactogenicity on an individual's physical functioning (PF) and QoL, the study will compare subject questionnaire responses made during two periods, i.e., pre-vaccination and post-vaccination. The difference will be considered to be the effect of vaccination and reactogenicity on the PF and QoL. To characterize the study population and determine if frailty may influence reactogenicity and consequently the impact on QoL scores, the subjects' frailty status will be assessed at the first inclusion visit. In addition to the SF-36 and EQ-5D questionnaires, a more complete characterization of the reactogenicity of the vaccine will be made by including a detailed collection of the use of healthcare resources and the occurrence of symptoms through diary card data collection. Impact on days of work loss, both for the subject or for a caregiver, as applicable, will also be assessed.

Note that as a result of internal change in data standards terminology, the study data collected was converted to cDISC and the statistical analysis plan was amended accordingly. "Day 0" in the study design was replaced by "Day 1"; consequently, "Day n" was replaced by "Day n+1". Thus, the timeframes (Day 0, Day n) of Outcome Measures described in this study record are different to that denoted in the full protocol document posted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the questionnaires and diary cards).
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* A male or female aged ≥ 50 YOA at the time of consent.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * For this study population, non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Any condition which, in the judgment of the investigator, would make intramuscular (IM) injection unsafe.
* Use or planned use of any investigational or non-registered product (drug or vaccine) other than the study vaccine or current participation or planned concurrent participation in another clinical study, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device) during the period starting 30 days before the first dose of study vaccine and the study end.
* Use or anticipated use of immunosuppressants or other immune-modifying drugs during the period starting 180 days prior to study start and during the whole study period. This includes chronic administration of corticosteroids (> 14 consecutive days of prednisone at a dose of ≥ 20 mg/day [or equivalent]), long-acting immune-modifying agents (e.g., infliximab) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders). Inhaled, topical and intra-articular corticosteroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, human immunodeficiency virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* Administration of immunoglobulins and/or any blood products in the period starting 90 days preceding the first dose of study vaccine or planned administration during the study period.
* Administration or planned administration of a live vaccine in the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine, or, administration or planned administration of a non-replicating vaccine in the period starting 15 days prior to and ending 14 days after either dose of study vaccine.
* Previous or planned administration of a vaccine against HZ (including an investigational or non-registered vaccine) other than the study vaccine, during the entire study period.
* History of HZ.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Pregnant or lactating female.
* Significant underlying illness requiring medications that might confound the evaluation of general/ local AEs, or in the opinion of the investigator, would be expected to prevent completion of the study.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (10):
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Norfolk, Virginia

REFERENCES:
- [Derived] Schmader KE, Levin MJ, Grupping K, Matthews S, Butuk D, Chen M, Idrissi ME, Fissette LA, Fogarty C, Hartley P, Klein NP, Nevarez M, Uusinarkaus K, Oostvogels L, Curran D. The Impact of Reactogenicity After the First Dose of Recombinant Zoster Vaccine on the Physical Functioning and Quality of Life of Older Adults: An Open-Label, Phase III Trial. J Gerontol A Biol Sci Med Sci. 2019 Jul 12;74(8):1217-1224. doi: 10.1093/gerona/gly218. PMID 30256905

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 404 subjects were enrolled in the study. However,1 subject was considered not eligible per the exclusion criteria (had previously received a Zoster vaccine) & 2 subjects were not vaccinated due to voluntary consent withdrawal.Hence,401 subjects were considered to have started the study & administered the first study vaccine (Exposed Set)
Groups:
- GSK1437173A Group: Subjects ≥ 50 years of age who received two doses of the GSK1437173A vaccine (first dose given at Month 0 and second dose given 2 months later) in this study.
Period: Overall Study
Arm/Group | GSK1437173A Group
Started | 401
Completed | 387
Not Completed | 14
Not completed — Withdrawal based on medical judgement | 1
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235
  Male | 166
Race/Ethnicity, Customized [Number; unit: Participants]
  African Heritage/African American | 48
  American Indian or Alaskan Native | 7
  Asian - East Asian Heritage | 2
  Asian - South East Asian Heritage | 1
  Other | 4
  White - Arabic / North African Heritage | 7
  White - Caucasian / European Heritage | 332

OUTCOME MEASURES:

1. Primary Outcome: Change in the Short Form 36-item-health Survey (SF36) Physical Functioning (PF) From Baseline Score to Mean Score After First Dose
Description: Descriptive analysis of the mean and standard deviation (SD) of the change from baseline of the SF-36 physical functioning (PF) score pre- and post dose 1 overall. Changes in the score were measured as Baseline versus mean score over the period Day 2 to Day 8 after first vaccination. Baseline for dose 1 is defined as the mean of the assessments at Day -7 and Day 1. The post-vaccination completion of SF-36 questionnaires brought home by the subjects were Days 2 to 7, with Day 8 to be filled in at the site. The SF-36 scale scores are constructed following the summated ratings of the questions and standardized SF-36 scoring algorithm. Scores range from 0 to 100, with a higher score representing a higher level of functioning.
Time Frame: From Baseline at Day -7 to Day 8 after first dose
Population: The analysis was performed on the Exposed Set, which included all vaccinated subjects with respect to the vaccine actually administered.
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 400
Score units | 1.9 (10.44)

2. Secondary Outcome: Change in Mean SF-36 PF Scale Scores From Baseline Score to Mean Score After Second Dose
Description: Descriptive analysis of the mean and standard deviation of the change from baseline of the SF-36 PF scale score pre and post dose 2 overall. Changes in the score were measured as Baseline versus mean score over the period Day 2 to Day 8 after second vaccination. For dose 2 baseline is defined as the mean of the three assessments at Day -7, Day 1 and Day 61 (Day 1 for dose 2). The post-vaccination completion of SF-36 questionnaires brought home by the subjects were on Day 2 to Day 7, with Day 8 to be filled in at the site. The SF-36 scale scores are constructed following the summated ratings of the questions and standardized SF-36 scoring algorithm. Scores range from 0 to 100, with a higher score representing a higher level of functioning.
Time Frame: From Day -7 to first dose until Day 8 after second dose (equivalent to study Days -7 to 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 389
Score units | -0.4 (10.38)

3. Secondary Outcome: Change in Mean SF-36 PF Single Item Scores After First Dose
Description: Descriptive analysis of the change in mean SF-36 PF single item score from baseline. Changes in the score were measured as Baseline versus mean score over the period Day 2 to Day 8 after the first vaccination. Baseline for dose 1 is defined as the mean of the assessments at Day -7 and Day 1. The post-vaccination completion of SF-36 questionnaires brought home by the subjects were Days 2 to 7, with Day 8 to be filled in at the site. The SF-36 scale scores are constructed following the summated ratings of the questions and standardized SF-36 scoring algorithm. Scores range from 0 to 100, with a higher score representing a higher level of functioning. Among items are vigorous activities (running, lifting heavy objects, participating in strenuous sports), moderate activities (moving a table, pushing a vaccum cleaner, bowling, or playing golf) and others, described in the categories below.
Time Frame: From Baseline at Day -7 to Day 8 after first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 400
Score units
  Vigorous activites | 6.8 (26.26)
  Moderate activites | 1.5 (16.76)
  Lifting or carrying groceries | 1.5 (13.84)
  Climbing several flights | 0.7 (17.77)
  Climbing one flight | 0.5 (16.26)
  Bending, kneeling or stooping | 5.8 (19.86)
  Walking more than a mile | -0.2 (19.28)
  Walking several hundred yards | -0.1 (16.66)
  Walking one hundred yards | 1.8 (15.11)
  Bathing or dressing himself/herself | 0.9 (11.35)

4. Secondary Outcome: Change in Mean SF-36 PF Single Item Scores After Second Dose
Description: Descriptive analysis of the change in mean SF-36 PF single item score from baseline. Baseline versus mean score over the period Day 2 to Day 8 after each vaccination. For dose 2 baseline is defined as the mean of the three assessments at Day -7, Day 1 and Day 61 (equivalent to Day 1 for dose 2) The post-vaccination completion of SF-36 questionnaires brought home by the subjects were on Day 2 to Day 7, with Day 8 to be filled in at the site. The SF-36 scale scores are constructed following the summated ratings of the questions and standardized SF-36 scoring algorithm. Scores range from 0 to 100, with a higher score representing a higher level of functioning. Among items are vigorous activities (running, lifting heavy objects, participating in strenuous sports), moderate activities (moving a table, pushing a vaccum cleaner, bowling, or playing golf) and others, described in the categories below.
Time Frame: From Day -7 to first dose until Day 8 after second dose (equivalent to study Days -7 to 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 389
Score units
  Vigorous activities | 2.6 (22.58)
  Moderate activities | -1.2 (16.82)
  Carrying groceries | -0.2 (13.05)
  Climbing several flights | -3.7 (18.76)
  Climbing one flight | -1.6 (16.09)
  Bending or kneeling | 3.9 (19.32)
  Walking more than mile | -2.3 (17.77)
  Walking several 100 yards | -2.0 (15.30)
  Walking 100 Yards | -0.1 (13.48)
  Bathing/dressing self | 1.0 (12.01)

5. Secondary Outcome: Change in SF-36 Role Physical Scores After First Dose
Description: Descriptive analysis. SF-36 Role physical scores change was measured from baseline score. Baseline versus mean score on Day 8 after first vaccination. Baseline for dose 1 is defined as the mean of the assessments at Day -7 and Day 1. The post-vaccination completion of SF-36 questionnaires brought home by the subjects were on Day 2 to Day 7, with Day 8 to be filled in at the site. The SF-36 scale scores are constructed following the summated ratings of the questions and standardized SF-36 scoring algorithm. Scores range from 0 to 100, with a higher score representing a higher level of functioning.
Time Frame: From Baseline at Day -7 to Day 8 after first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 286
Score units | 1.4 (14.97)

6. Secondary Outcome: Change in SF-36 Role Physical Scores After Second Dose
Description: Descriptive analysis. SF-36 Role Physical scores change was measured from baseline score. Changes in the score were measured as Baseline versus Day 8 score after the second vaccination. For dose 2 baseline is defined as the mean of the three assessments at Day -7, Day 1 and Day 61 (equivalent to Day 1 for dose 2) The post-vaccination completion of SF-36 questionnaires brought home by the subjects were on Day 2 to Day 7, with Day 8 to be filled in at the site. The SF-36 scale scores are constructed following the summated ratings of the questions and standardized SF-36 scoring algorithm. Scores range from 0 to 100, with a higher score representing a higher level of functioning.
Time Frame: From Day -7 to first dose until Day 8 after second dose (equivalent to study Days -7 to 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 291
Score units | -1.8 (16.40)

7. Secondary Outcome: Change in Quality-adjusted Life Year (QALY) After First Dose
Description: Descriptive analysis. QALY estimation is done from baseline score, based on EQ-5D questionnaires. Baseline versus combined score over the period Day 2 to Day 8 after each vaccination. Baseline for dose 1 is defined as the mean of the assessments at Day -7 and Day 1. The post-vaccination completion of EQ-5D questionnaires brought home by the subjects were on Day 2 to Day 7, with Day 8 to be filled in at the site. The EQ-5D is a generic measure of health status that provides a simple description profile based on 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, which are used to generate the EQ-5D index utility score. The EQ-5D index utility score ranges from 0 (worst health state) to 1 (perfect health state); 1 reflects the best outcome.
Time Frame: From Baseline at Day -7 to Day 8 after first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 399
Score units | 0.1829 (0.55551)

8. Secondary Outcome: Change in QALY After Second Dose
Description: Descriptive analysis. QALY estimation is done from baseline score, based on EQ-5D questionnaires. Baseline versus combined score over the period Day 2 to Day 8 after each vaccination. For dose 2 baseline is defined as the mean of the three assessments at Day -7, Day 1 and Day 61 (equivalent to Day 1 for dose 2) The post-vaccination completion of SF-36 and EQ-5D questionnaires brought home by the subjects were on Day 2 to Day 7, with Day 8 to be filled in at the site. The EQ-5D is a generic measure of health status that provides a simple description profile based on 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5 items are combined to generate health profiles (e.g. 1-no problem/no symptom) and profiles are subsequently converted to a continuous single index utility score (higher scores represent a better quality of life).
Time Frame: From Day -7 to first dose until Day 8 after second dose (equivalent to study Days -7 to 68)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score units
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 388
Score units | 0.1128 (0.52000)

9. Secondary Outcome: Number of Reactogenicity-triggered Medically Attended Visits After First Dose
Description: Medical attention and health resource utilization triggered by frequency of reactogenicity events. Healthcare resources included staff involved in the following activities: telephone calls, visit to general practitioner, visit to specialist, visit to emergency room and hospitalizations.
Time Frame: From Day 1 to Day 7 after first dose
Population: as for outcome 1
Measure: Number; unit: Visits
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 401
Visits
  Attended by Telephone Call | 2
  Attended by General Practicioner | 1
  Attended by Specialist | 0
  Attended by Emergency Room | 0
  Attended by Hospitalization | 0

10. Secondary Outcome: Number of Reactogenicity-triggered Medically Attended Visits After Second Dose
Description: as for outcome 9
Time Frame: From Day 1 to Day 7 after second dose
Population: as for outcome 1
Measure: Number; unit: Visits
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 391
Visits
  Attended by Telephone Call | 4
  Attended by General Practitioner | 1
  Attended by Specialist | 0
  Attended by Emergency Room | 0
  Attended by Hospitalization | 0

11. Secondary Outcome: Days of Work Loss for Subjects After First Dose
Description: Descriptive analysis. Estimation of work loss due to any reaction related to the study vaccine for subjects, expressed in days.
Time Frame: From Day 1 to Day 7 after first dose
Population: The analysis was performed on the total number of subjects who reported work loss after the first vaccination and were part of the exposed set, which included all vaccinated subjects with respect to the vaccine actually administered
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 5
Days | 1.3 (1.0)

12. Secondary Outcome: Days of Work Loss for Subjects After Second Dose
Description: as for outcome 11
Time Frame: From Day 1 to Day 7 after second dose
Population: The analysis was performed on the total number of subjects who reported work loss after the second dose and were part of the exposed set, which included all vaccinated subjects with respect to the vaccine actually administered
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 13
Days | 1.1 (0.4)

13. Secondary Outcome: Days of Work Loss for Non-dedicated Caregivers After First Dose
Description: Descriptive analysis. Estimation of work loss of non-dedicated caregivers expressed in days.Data was not reported for this outcome measure as there was no work loss among the non-dedicated caregivers
Time Frame: From Day 1 to Day 7 after first dose
Population: The analysis was performed on the total number of non-dedicated caregivers who reported work loss after the first dose and were part of the exposed set, which included all vaccinated subjects with respect to the vaccine actually administered
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 0

14. Secondary Outcome: Days of Work Loss for Non-dedicated Caregivers After Second Dose
Description: Descriptive analysis. Estimation of work loss due to any reaction related to the study vaccine for non-dedicated caregivers, expressed in days. Data was not reported for this outcome measure as there was no work loss among the non-dedicated caregivers
Time Frame: From Day 1 to Day 7 after second dose
Population: The analysis was performed on the total number of non-dedicated caregivers who reported work loss after second dose and were a part of the exposed set, which included all vaccinated subjects with respect to the vaccine actually administered.
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 0

15. Secondary Outcome: Days of Extra Work for Dedicated Caregivers After First Dose
Description: Descriptive analysis. Estimation of extra work for dedicated caregivers. Data was not reported for this outcome measure as there was no extra work for the dedicated caregivers
Time Frame: From Day 1 to Day 7 after first dose
Population: The analysis was performed on the total number of dedicated caregivers who reported extra work after the first dose and were part of the exposed set, which included all vaccinated subjects with respect to the vaccine actually administered.
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 0

16. Secondary Outcome: Days of Extra Work for Dedicated Caregivers After Second Dose
Description: Descriptive analysis. Estimation of extra work for dedicated caregivers, expressed in days. Data was not reported for this outcome measure as there was no extra work for the dedicated caregivers
Time Frame: From Day 1 to Day 7 after second dose
Population: The analysis was performed on the total number of dedicated caregivers who reported extra work after second dose and were part of the exposed Set, which included all vaccinated subjects with respect to the vaccine actually administered.
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms After First Dose
Description: Assessed solicited local symptoms were pain, erythema and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 erythema/swelling =erythema/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after first dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 400
Participants
  Any Pain | 310
  Grade 3 Pain | 16
  Any Erythema | 92
  Grade 3 Erythema | 6
  Any Swelling | 53
  Grade 3 swelling | 3

18. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms After Second Dose
Description: Assessed solicited local symptoms were pain, erythema and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 erythema/swelling=erythema/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after second dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 389
Participants
  Any Erythema | 87
  Grade 3 Erythema | 7
  Any Pain | 292
  Grade 3 Pain | 21
  Any Swelling | 54
  Grade 3 Swelling | 3

19. Secondary Outcome: Number of Days With Solicited Local Symptoms After First Dose
Description: Assessed solicited local symptoms were pain, erythema and swelling.
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after first dose.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 400
Days
  Pain: number analyzed (Participants) | 310
  Pain | 3 [2 to 4]
  Erythema: number analyzed (Participants) | 92
  Erythema | 2 [2 to 4]
  Swelling: number analyzed (Participants) | 53
  Swelling | 2 [2 to 4]

20. Secondary Outcome: Number of Days With Solicited Local Symptoms After Second Dose
Description: Assessed solicited local symptoms were pain, erythema and swelling.
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after second dose.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 292
Days
  Pain | 2.5 [2 to 3]
  Erythema: number analyzed (Participants) | 87
  Erythema | 3.0 [2 to 4]
  Swelling: number analyzed (Participants) | 54
  Swelling | 3.0 [1 to 4]

21. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms After First Dose
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia, shivering and temperature [defined as oral, axillary or tympanic temperature equal to or above (≥)37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal everyday activities. Grade 3 temperature=temperature≥39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after first dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 400
Participants
  Any Fatigue | 134
  Grade 3 Fatigue | 13
  Related Fatigue | 120
  Any Gastrointestinal symptoms | 53
  Grade 3 Gastrointestinal symptoms | 4
  Related Gastrointestinal symptoms | 40
  Any Headache | 113
  Grade 3 Headache | 11
  Related Headache | 98
  Any Myalgia | 107
  Grade 3 Myalgia | 8
  Related Myalgia | 100
  Any Shivering | 50
  Grade 3 Shivering | 3
  Related Shivering | 48
  Any Temperature (oral route) | 37
  Grade 3 Temperature(≥39.0 °C) | 0
  Related Temperature | 34

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms After Second Dose
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia, shivering and temperature [defined as oral, axillary, tympanic temperature ≥ 37.5 °C]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = temperature≥39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after second dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 389
Participants
  Any Fatigue | 180
  Grade 3 Fatigue | 27
  Related Fatigue | 172
  Any Gastrointestinal symptoms | 53
  Grade 3 Gastrointestinal symptoms | 4
  Related Gastrointestinal symptoms | 44
  Any Headache | 146
  Grade 3 Headache | 11
  Related Headache | 127
  Any Myalgia | 128
  Grade 3 Myalgia | 16
  Related Myalgia | 121
  Any Shivering | 97
  Grade 3 Shivering | 14
  Related Shivering | 86
  Any Temperature (oral route) | 69
  Grade 3 Temperature(≥39.0 °C) | 1
  Related Temperature | 64

23. Secondary Outcome: Number of Days With Solicited General Symptoms After First Dose
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia, shivering and temperature [defined as oral, axillary or tympanic temperature equal to or above (≥)37.5 degrees Celsius (°C)].
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after first dose.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 400
Days
  Fatigue: number analyzed (Participants) | 134
  Fatigue | 2 [1 to 3]
  Gastrointestinal symptoms: number analyzed (Participants) | 53
  Gastrointestinal symptoms | 1 [1 to 3]
  Headache: number analyzed (Participants) | 113
  Headache | 2 [1 to 3]
  Myalgia: number analyzed (Participants) | 107
  Myalgia | 2 [1 to 3]
  Shivering: number analyzed (Participants) | 50
  Shivering | 1 [1 to 2]
  Temperature: number analyzed (Participants) | 37
  Temperature | 1 [1 to 2]

24. Secondary Outcome: Number of Days With Solicited General Symptoms After Second Dose
Description: as for outcome 23
Time Frame: During a 7-day follow-up period (Day 1 to Day 7) after second dose.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 180
Days
  Fatigue | 2.0 [1 to 3]
  Gastrointestinal symptoms: number analyzed (Participants) | 53
  Gastrointestinal symptoms | 2.0 [1 to 3]
  Headache: number analyzed (Participants) | 146
  Headache | 1.5 [1 to 2]
  Myalgia: number analyzed (Participants) | 128
  Myalgia | 2.0 [1 to 3]
  Shivering: number analyzed (Participants) | 97
  Shivering | 1.0 [1 to 2]
  Temperature: number analyzed (Participants) | 69
  Temperature | 1.0 [1 to 1]

25. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
  Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During a 30-day follow-up period (Day 1 to Day 30) after any vaccination (across doses).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 401
Participants
  Any unsolicited adverse event | 127
  Grade 3 unsolicited adverse events | 25
  Related unsolicited adverse events | 29

26. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs) During the Entire Study Period
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 1 to study end at Month 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 401
Participants
  Any SAEs | 14
  Related SAEs | 0

27. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 1 to study end at Month 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group
Number analyzed (Participants) | 401
Participants
  Any pIMDs | 2
  Related pIMDs | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general adverse events: Day 1 to 7 after each vaccination. Unsolicited adverse events: From Day 1-30 after each vaccination. SAEs: From Day 1 to study completion (month 14).
Arm/Group | GSK1437173A Group
All-Cause Mortality (participants affected / at risk) | 2/401
Serious Adverse Events (participants affected / at risk) | 14/401
Other Adverse Events (participants affected / at risk) | 370/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=401)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=401)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) — Unsolicited symptoms
Atrial fibrilation (Cardiac disorders) | 1 (1) — Unsolicited symptoms
Vertigo (Ear and labyrinth disorders) | 2 (2) — Unsolicited symptoms
Conjunctivitis allergic (Eye disorders) | 1 (1) — Unsolicited symptoms
Eye irritation (Eye disorders) | 1 (1) — Unsolicited symptoms
Eye pain (Eye disorders) | 2 (2) — Unsolicited symptoms
Keratitis (Eye disorders) | 1 (1) — Unsolicited symptoms
Constipation (Gastrointestinal disorders) | 1 (1) — Unsolicited symptoms
Diarrhoea (Gastrointestinal disorders) | 1 (1) — Unsolicited symptoms
Gastrointestinal disorder (Gastrointestinal disorders) | 88 (107) — Unsolicited symptoms
Haematochezia (Gastrointestinal disorders) | 1 (1) — Unsolicited symptoms
Haemorrhoids (Gastrointestinal disorders) | 1 (1) — Unsolicited symptoms
Nausea (Gastrointestinal disorders) | 4 (4) — Unsolicited symptoms
Toothache (Gastrointestinal disorders) | 1 (1) — Unsolicited symptoms
Vomiting (Gastrointestinal disorders) | 3 (3) — Unsolicited symptoms
Application site erythema (General disorders) | 1 (1) — Unsolicited symptoms
Application site hyperaesthesia (General disorders) | 1 (1) — Unsolicited symptoms
Chills (General disorders) | 115 (148) — Unsolicited symptoms
Fatigue (General disorders) | 227 (315) — Unsolicited symptoms
Feeling cold (General disorders) | 1 (1) — Unsolicited symptoms
Ill-defined disorder (General disorders) | 1 (1) — Unsolicited symptoms
Inflammation (General disorders) | 1 (1) — Unsolicited symptoms
Injection site bruising (General disorders) | 2 (2) — Unsolicited symptoms
injection site erythema (General disorders) | 125 (180) — Unsolicited symptoms
Injection site pain (General disorders) | 341 (603) — Unsolicited symptoms
Injection site pruritus (General disorders) | 8 (9) — Unsolicited symptoms
Injection site warmth (General disorders) | 1 (1) — Unsolicited symptoms
Malaise (General disorders) | 2 (2) — Unsolicited symptoms
Oedema peripheral (General disorders) | 1 (1) — Unsolicited symptoms
Pain (General disorders) | 2 (2) — Unsolicited symptoms
Peripheral swelling (General disorders) | 2 (2) — Unsolicited symptoms
Pyrexia (General disorders) | 88 (107) — Unsolicited symptoms
Seasonal allergy (Immune system disorders) | 1 (1) — Unsolicited symptoms
Bronchitis (Infections and infestations) | 5 (5) — Unsolicited symptoms
Cystitis (Infections and infestations) | 2 (2) — Unsolicited symptoms
Eye infection staphilococcal (Infections and infestations) | 1 (1) — Unsolicited symptoms
Fungal infection (Infections and infestations) | 1 (1) — Unsolicited symptoms
Gastroenteritis viral (Infections and infestations) | 1 (1) — Unsolicited symptoms
Gastrointestinal viral infection (Infections and infestations) | 1 (1) — Unsolicited symptoms
Groin abcess (Infections and infestations) | 1 (1) — Unsolicited symptoms
Nasopharyngithis (Infections and infestations) | 10 (10) — Unsolicited symptoms
Oral herpes (Infections and infestations) | 4 (4) — Unsolicited symptoms
Pneumonia (Infections and infestations) | 1 (1) — Unsolicited symptoms
Rhinitis (Infections and infestations) | 1 (1) — Unsolicited symptoms
Sinusitis (Infections and infestations) | 6 (6) — Unsolicited symptoms
Tooth abcess (Infections and infestations) | 2 (2) — Unsolicited symptoms
Tooth infection (Infections and infestations) | 1 (1) — Unsolicited symptoms
Upper respiratory tract infection (Infections and infestations) | 8 (8) — Unsolicited symptoms
Urinary tract infection (Infections and infestations) | 4 (4) — Unsolicited symptoms
Viral infection (Infections and infestations) | 2 (2) — Unsolicited symptoms
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Fall (Injury, poisoning and procedural complications) | 2 (2) — Unsolicited symptoms
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 (1) — Unsolicited symptoms
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) — Unsolicited symptoms
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) — Unsolicited symptoms
Gout (Metabolism and nutrition disorders) | 1 (2) — Unsolicited symptoms
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — Unsolicited symptoms
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) — Unsolicited symptoms
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unsolicited symptoms
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) — Unsolicited symptoms
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) — Unsolicited symptoms
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 (2) — Unsolicited symptoms
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Unsolicited symptoms
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (4) — Unsolicited symptoms
Myalgia (Musculoskeletal and connective tissue disorders) | 169 (238) — Unsolicited symptoms
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) — Unsolicited symptoms
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unsolicited symptoms
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) — Unsolicited symptoms
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) — Unsolicited symptoms
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unsolicited symptoms
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Unsolicited symptoms
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unsolicited symptoms
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Unsolicited symptoms
Dizziness (Nervous system disorders) | 5 (5) — Unsolicited symptoms
Headache (Nervous system disorders) | 189 (268) — Unsolicited symptoms
Hypoaesthesia (Nervous system disorders) | 3 (4) — Unsolicited symptoms
Lethargy (Nervous system disorders) | 3 (3) — Unsolicited symptoms
Migraine (Nervous system disorders) | 1 (1) — Unsolicited symptoms
Paraesthesia (Nervous system disorders) | 2 (2) — Unsolicited symptoms
Sciatica (Nervous system disorders) | 2 (2) — Unsolicited symptoms
Sinus headache (Nervous system disorders) | 1 (1) — Unsolicited symptoms
Anxiety (Psychiatric disorders) | 1 (1) — Unsolicited symptoms
Insomnia (Psychiatric disorders) | 2 (2) — Unsolicited symptoms
Panic attack (Psychiatric disorders) | 1 (1) — Unsolicited symptoms
Stress (Psychiatric disorders) | 1 (1) — Unsolicited symptoms
Nephrolithiasis (Renal and urinary disorders) | 1 (1) — Unsolicited symptoms
Urinary tract disorder (Renal and urinary disorders) | 1 (1) — Unsolicited symptoms
Urine odour abnormal (Renal and urinary disorders) | 1 (1) — Unsolicited symptoms
Pelvic pain (Reproductive system and breast disorders) | 1 (1) — Unsolicited symptoms
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unsolicited symptoms
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) — Unsolicited symptoms
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Unsolicited symptoms
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Unsolicited symptoms
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unsolicited symptoms
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Unsolicited symptoms
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unsolicited symptoms
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — Unsolicited symptoms
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) — Unsolicited symptoms
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) — Unsolicited symptoms
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) — Unsolicited symptoms
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — Unsolicited symptoms
Sinus operation (Surgical and medical procedures) | 1 (1) — Unsolicited symptoms
Flushing (Vascular disorders) | 1 (1) — Unsolicited symptoms
Injection site swelling (General disorders) | 78 (107)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT02979639/SAP_000.pdf
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT02979639/Prot_001.pdf